CLINICAL TRIAL: NCT06684977
Title: Virtual Reality and Post-Traumatic Stress - Exploring the Feasibility and Acceptability of Low-Cost Virtual Reality and 360 Video to Treat Post Traumatic Stress Disorder
Brief Title: Virtual Reality and Post Traumatic Stress
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: South Eastern Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Dr Paul Best, Principle Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS Project ID - 325495
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; Trauma; Virtual Reality; Mental Health
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment As Usual (Active Comparator): (N=5) as a control group who will only receive TF-CBT.
- 360 Video (Experimental): (N=5) to use 360° Video alongside standard TF-CBT.
- VR Photoscan (Experimental): (N=5) to use VR Photo Scan alongside standard TF-CBT.

INTERVENTIONS:
Behavioral: 360 Video — 360° Video consists of video recordings, made with a camera to simultaneously capture and combine scenes in a 360 degrees perspective such as Instant Google Street View Instant Google Street View (instantstreetview.com). When uploaded to a VR headset, 360° videos may provide a more cost-effective method for rapidly creating virtual environments in which users can experience a sense of immersion and the viewer can control and change the viewing angle at any stage through head movement. While photorealism may be superior, this option is known to be less interactive as the viewer can't move or walk around within the virtual space. In addition, the landscape and imagery may have been changed or developed meaning the recordings captured do not match the traumatic memory. Despite these limitations, the use of 360° video has been trialled in clinical mental health settings showing positive outcomes for both user and clinician.
Behavioral: VR Photoscan — VR Photoscan creates immersive virtual environments by transforming real-world imagery into detailed 3D models. Using high-resolution images captured from a smartphone, these images are processed in 3D graphics software to sculpt realistic virtual scenes. The resulting 3D models are imported into a game engine, adding VR functionality, allowing users to navigate freely with six degrees of freedom. Interactive content, such as animated cars and people, can be added in real-time, while menu systems guide users through the experience. Environmental factors like lighting, weather, and time of day can be adjusted to simulate real conditions. Spatial 360° audio enhances immersion, providing sounds from various directions. This VR environment creation process is efficient and cost-effective, requiring no specialised equipment, and ensuring high-quality immersive experiences at minimal production time and cost.
Behavioral: Standard TF-CBT — Ehlers and Clark's model follows the general style of reliving (recommended by NICE) suggested by Foa and Rothbaum with some fluidity and in vivo exposure (i.e., trauma site visit). During the treatment process of reliving, clients are asked to close their eyes and intentionally recall the traumatic memories, i.e., relive the trauma in their mind in detail and narrate their experience in present tense, including recalling images, sensory experiences, thoughts, and feelings. VR-based PTSD treatments can promote emotional engagement and the process of trauma via providing visual, auditory, and haptic sensory cues.

SUMMARY:
Northern Ireland has a legacy of trauma-related mental health problems and a higher estimated prevalence of post-traumatic stress disorder (PTSD) than other comparable post-civil conflict societies. Trauma-Focused Cognitive Behavioural Therapy (TF-CBT) is an effective treatment for PTSD and is currently recommended by the National Institute For Health and Social Care Excellence (NICE) as the first line of clinical treatment. During therapy, clients with PTSD revisit the trauma memory to process what has occurred. This technique is known as Imaginal Exposure (IE) which can be a difficult process. Clients can be highly avoidant and emotionally distant from trauma memories, making it challenging to engage with the exposure process. When trauma has occurred several decades previously, traumatic memories may be difficult to access, resulting in poor treatment outcomes.

Technology such as Virtual Reality (VR) can aid this process, as patients can enter a world that exposes them to the traumatic memory in a controlled therapeutic way which has shown to be effective in the treatment of PTSD. VR is yet to be used in routine clinical settings. The investigators are proposing to create low-cost VR environments via 360° video and a new process called VR Photoscan, which will allow a clinical setting to use this beneficial tool to support patients who are receiving TF-CBT to treat PTSD.

This is a three-arm intervention feasibility study using a mixed methods evaluation framework designed to explore the acceptability of low-cost VR as an adjunct within existing TF-CBT therapy.

Participants will be split into 3 groups of 5:

Group one (N=5) to use 360° Video alongside standard TF-CBT. Group two (N=5) to use VR Photo Scan alongside standard TF-CBT. Group three (N=5) is a control group that will only receive TF-CBT.

The individuals selected for the technological interventions will be offered the opportunity of a personalized 360° video / VR Photoscan environment to aid their therapy session. Pre and post-measures will be collected from participants and semi-structured interviews will be held with participants at the end of their therapy and with the clinicians who have delivered the intervention. This protocol aims to investigate the potential of low-cost VR technology in supporting PTSD treatment, addressing both the practical and theoretical challenges of immersive trauma therapy. By examining the feasibility of 360° video and VR Photoscan, the study hopes to contribute valuable insights into VR's applicability in clinical mental health settings.

DETAILED DESCRIPTION:
Background Northern Ireland is a country that has recently emerged from around 30 years of civil conflict that has resulted in the deaths of over 3500 people. This period known colloquially as 'The Troubles' has resulted in a legacy of trauma-related mental health problems and has a higher estimated prevalence of Post-Traumatic Stress Disorder (PTSD) than any other comparable country that has experienced civil conflict. This has resulted in an estimated 39% of the population experiencing (directly or indirectly) a conflict-related 'event'. PTSD has an estimated prevalence of 3.6% in the general world population and a disproportionately high prevalence of 5.1% among the Northern Ireland population.

Trauma-Focused Cognitive Behavioural Therapy (TF-CBT) has been demonstrated to be an effective treatment for PTSD evolved from the Ehlers and Clark Cognitive Model of persistent PTSD. The evidence-based treatment of non-conflict related trauma such as sexual assault, and road traffic accidents has highlighted the effectiveness and common acceptance of TF-CBT and is currently recommended by the NICE as the first line of clinical treatment for PTSD. TF-CBT for individuals in Northern Ireland suffering from PTSD which has arisen from acts of terrorism and civil conflict has added to the emergent evidence base as a successful therapeutic intervention.

The model, Ehlers & Clark, suggests that PTSD can develop if the patient continues to feel a sense of current threat after the trauma has ended, which can lead to further dysfunctional behaviors and feelings, even after the event has taken place. During the course of therapy, clients with PTSD revisit the trauma memory in order to fully process what has occurred. This technique is known as Imaginal Exposure (IE) via Reliving and whilst shown to be effective, IE can be a difficult process for clients given the associated, somatic and cognitive symptoms that it incurs. People diagnosed with PTSD can be highly avoidant and emotionally distant from trauma memories, meaning they find it challenging to engage with the exposure process. In addition, when trauma has occurred several decades previously, the trauma memory may be difficult to access or may have lost detail resulting in poor treatment outcomes.

Given the role of imaginal techniques within PTSD treatment, a growing number of studies have explored the use of immersive technology such as Virtual Reality (VR) to support this process. VR is no longer a futuristic concept and headsets are readily accessible, being used in many households for entertainment purposes. Currently, there are many ways to create a virtual world and if used correctly can be therapeutically helpful to patients and clinicians. VR can generate environments such as social settings or classrooms that essentially simulate real or imagined worlds to meet the specific clinical requirements of the patient in therapy. Through the use of VR, patients can enter a world in which they are exposed to a traumatic memory in a controlled therapeutic way, and, as a result, has been shown to be effective in the treatment of PTSD patients across a number of settings such as military combat, terrorist attacks, and road traffic accidents. Specific to the military, in 2003, due to the deployments to Afghanistan and Iraq there was an increase in combat-related PTSD which the United States recognised the need to advance in evidence-based treatments to address these complexities. Despite these successes, there is yet to be a widespread adoption of VR-based interventions for PTSD in routine clinical settings. Potential barriers are hypothesized to occur due to the idiosyncratic nature of the trauma memory, which requires the recreation of a personalized environment and thus has significant cost implications. Another barrier may be due to the acceptability or lack thereof of these new technologies among clinicians.

Theoretical Framework

The clinical presentation of PTSD is idiosyncratic; with specific symptoms experienced differing from individual to individual. Unwanted, intrusive, and involuntary distressing memories of the traumatic event are a core symptom of PTSD. Most successful treatment protocols for PTSD focus on the patient's memory of the traumatic event and its meaning. Therefore, a range of interventions have been developed to reduce the stress associated with these memories. Such interventions include Prolonged Exposure (PE), imaginal reliving of the trauma, and cognitive interventions to support the elaboration of traumatic memory to link with autobiographical memories. For this study, Ehlers and Clark's Cognitive Model of Persistent PTSD was used as a framework to develop the current treatment protocol.

In their cognitive model, they posit that chronic PTSD develops because individuals engage in sensory processing of the event rather than processing the meaning and implications. This causes disturbance in autobiographical memory, i.e., episodic (personal memories including places, objects, events) and semantic memory (memories about general knowledge and facts). Subsequently, this prevents the processing of trauma memories. They also postulated that individuals who experience PTSD develop excessively negative appraisals in which the probability of risk of harm is overestimated, and the ability to cope with threat is underestimated. Such maladaptive cognitive errors/biases cause avoidance of threats and provide short-term relief. These include avoiding trauma-related stimuli, and remembering or suppressing unwanted trauma-related thoughts. However, in the long term, these activities maintain the sense of persistent threat as the coping strategies prevent negative appraisals from being corrected. Thus, the authors proposed that recalling the traumatic memories and updating them is the core of trauma treatment. Ehlers and Clark's model follows the general style of reliving (recommended by NICE) suggested by Foa and Rothbaum with some fluidity and in vivo exposure (i.e., trauma site visit). During the treatment process of reliving, clients are asked to close their eyes and intentionally recall the traumatic memories, i.e., relive the trauma in their mind in detail and narrate their experience in the present tense, including recalling images, sensory experiences, thoughts, and feelings. VR-based PTSD treatments can promote emotional engagement and the process of trauma by providing visual, auditory, and haptic sensory cues. The investigators posit that a similar effect can be achieved via the use of 360° video or VR Photoscan technologies.

This study seeks to address these barriers by implementing two acceptable but lower-cost alternatives to VR, namely (1) Immersive 360° Video and (2) VR Photoscan technology in a routine clinical setting in Northern Ireland.

Project Aim and Objectives This is a three-arm intervention feasibility study using a mixed methods evaluation framework designed to explore the acceptability of low-cost VR as an adjunct within existing TF-CBT therapy.

Objectives

1. To explore the user (clinician and patient) acceptability of 360° video and VR Photoscan within a routine mental healthcare setting.
2. To understand the factors surrounding the recruitment and retention of participants using 360° video and VR Photoscan within a routine mental healthcare setting.
3. To explore differences between participants receiving 360° video or VR Photoscan or treatment as usual (TAU) within a routine mental healthcare setting using a three-arm design.

Intervention Developments (See Arms and Interventions Section)

Methods

This is a three-arm intervention development study using a mixed methods evaluation framework designed to explore and refine the use of low-cost VR as an adjunct within existing TF-CBT therapy. The study will take place within the Regional Trauma Network based in the South-Eastern Trust (SET). This study of approximately 15 participants (N=15) selected from the waitlist will be screened for suitability of therapy to treat conflict-related PTSD. The participants will be split into three random N-5 groups.

Group one (N=5) to use 360° Video alongside standard TF-CBT. Group two (N=5) to use VR Photo Scan alongside standard TF-CBT. Group three (N=5) is a control group that will only receive TF-CBT. The individuals selected for the technological interventions will be offered the opportunity of a personalized 360° video / VR Photoscan environment to aid their therapy session.

It is preferred that the site trauma is suitable for the two arms of the study, but on the occasion that this is not possible, participants will be selected for each arm based on the accessibility of the trauma.

In line with the standard RTN OUTCOMES: MEASURES AGAINST STAGE OF THERAPY, each stage of treatment uses a choice of measures to collect data outcomes. (See the Outcome Measures section for more detail). Additionally, the co-researcher will hold semi-structured interviews to gather the views and experiences of the clinicians and clients once the intervention has ended.

Recruitment and Sampling

The target sample size is 15 participants (N-15). Recruitment is likely to take place in September 2023.

Numerous meetings have been held between the research team at QUB and the SET Regional Trauma Network to ensure the approach is refined and effective, ensuring the flow of the study and minimizing the additional workload for the clinicians involved. The Regional Trauma Network will be responsible for the recruitment under the lead of the Consultant Clinical Psychologist. Standard practice within the Regional Trauma Network is a four-stage RTN Flowchart in which during initial assessment baselines are collected and readiness and commitment for therapy are evaluated, at this stage a brief overview of the trauma location will be gathered and accessibility assessed for the purpose of the VR. It is amenable that both arms of the study are met however on the occasion this is not possible, participants will be selected based on suitability. A purposive sampling technique will gauge the service users' interest and suitability based on the exclusion and inclusion criteria of the study (See Eligibility section) which will be added to a series of questions within the RTN Screening Proforma. If clients show interest, the clinician will provide them with the Participants Information Sheet and the Consent Form. The decision to take part (or not) will not impact the service that they receive. As such, if the participant does not show interest in the study, they will remain on the standard treatment waitlist. Suitable participants will then be placed on a waitlist for the purpose of this study. As per the RTN Screening Proforma, the PIS will be disseminated to the GP alongside the Screening Outcome Letter to ensure the GP receives sufficient details on the study. The clinicians (N-5) identified to take part in the study are employed directly through SET are a Consultant Clinical Psychologist and four Psychological Therapists (Psychology, Nursing, and Social Work Core Professionals) trained in delivering TF-CBT. Each clinician will be trained in the use of both 360° video and VR Photoscan technologies. Patients will be screened with those referred earliest seen first. From the resultant list of consulting patients, they will be randomly allocated where possible to the three arms. A maximum of 5 patients per group will be assigned until all arms are full.

As per NICE guidelines standard treatment includes around 8-12 meetings and sessions at least approximately 60-90 minutes. As this study will be working with complex PTSD, therapy can run into 20+ sessions. The endpoint for data collection for this study will be after approximately 16-20 sessions

Randomization

Randomization will take place following registration and completion of baseline measures based on the acceptability of 360° video and VR Photoscan technology. Each participant will be assigned a unique individual number and a simple random sampling procedure will be performed using online software available at http://www.random.org. 3 sets of 5 unique numbers per set will be automated, ranging from 1 to 15. Each set will be allocated to either 360° video, VR Photoscan, or TAU groups. It is amenable that the index trauma location is accessible to be captured on both forms of technology to allow for randomization, however, on the occasion that the sample size cannot be met with this criteria, participants will be assigned into the arms of the study-based on the accessibility of the index trauma.

Intervention Delivery Protocol

360° video or VR Photoscan technology involves sculpting real-world imagery into a blank Virtual Reality canvas. This offers the user the benefits of increased photorealism while retaining the affordances offered by VR. To create these environments a simple 5-step protocol for each technology has been developed.

Once the 360° video or VR Photoscan environment has been uploaded, the clinician is able to use this as part of the imaginal exposure process contained within TF-CBT. All clinicians taking part in the study are qualified to deliver TF-CBT and have experience of treating PTSD using TF-CBT models. For this study and as per standard SET practice, the Ehlers and Clark Cognitive Model of PTSD is the chosen TF-CBT protocol. However, given the complex nature of PTSD, some variation of exposure dose, i.e., the number of VR sessions (and therefore the time spent in the 360° video or VR Photoscan environments) may occur across the sample. To minimize the impact of this, clinicians will use the 360° video or VR Photoscan environments as a substitute for imaginal exposure techniques during reliving sessions. In each session that VR is used, clinicians will be asked to complete a small check box that will monitor the length and number of sessions the VR is used.

Hardware

VR Photoscan environments will be captured via a photo on a smart mobile phone provided by clinicians or the co-researcher during the site visit. A 360° video camera will be provided by QUB and used by clinicians and the co-researcher to capture environments for the participants in this group. Alternatively, if required, Google Streetview can be accessed on the Oculus Quest headset for a 360° view of the site. The VR devices used for the intervention are Oculus Quest 2 headsets, provided for the duration of the study by QUB. This device is worn with T-straps holding it securely on the head, with a cable connected to the computer screen or the device can be wirelessly streamed to a phone or tablet. The screen will enable the clinician to view the participant's virtual environment. The VR headset will only be used during the sessions in which the exposure components of the TF-CBT protocol.

Statistical Methods and Analysis

Descriptive statistics, including means and standard deviations, will be calculated at each time point for each outcome. Recruitment (number of participants at the beginning of the study) and retention (numbers that complete the study, dropout) rates will be reported. The implementation of the treatment protocol will be described, and adverse events will be recorded and reported. Baseline measures will be provided to participants during the introductory sessions and outcomes will be analyzed and evaluated using the Statistical Package for Social Sciences, v26. As this is an intervention development study, no formal sample size calculations were conducted or required as part of the project aims/objectives. As such, the sample for the study has been based on practical considerations including cost and time available within the constraints of the allocated time. Confidence intervals will be provided along with any estimates, and any change in outcome scores between baseline (before the intervention), and post-intervention outcomes of both treatment groups using 360° video and VR Photoscan for further comparison and analysis. Adherence rates will also be analyzed and evaluated post-intervention. It is worth noting, however, that the study is not powered for significance testing so results will be interpreted with caution.

Qualitative data analysis will explore issues of acceptability (of the intervention); potential advantages and disadvantages of the intervention; practicalities of delivering the intervention; and the suitability of recruitment methods. A reflexive thematic analysis will be used for a theoretically flexible method following the six phases for collecting, analyzing, and reporting qualitative data - this will be supported by NVivo 14 software which the co-researcher will be fully trained on using.

Consent

The study will incorporate an opt-in consent procedure. Clinicians will be contacted via email with a study invitation and consent form to participate.

The clinical team will disseminate participants with an information sheet and obtain written consent from clients before baseline measures are given. This will include information and consent for the follow-up semi-structured interviews.

All participants will be made aware that withdrawing from the study will not affect their access to treatment within SET, or in any other organizations e.g., GP. Participants will be given an information sheet where they will be informed about the nature of the study, the potential benefits of participating, and how the data will be used. The information sheet will also explain that participation is voluntary and that participants' confidentiality will be protected throughout. Should participants consent to participate they will be provided with a consent form for completion. Participants will be allowed to address any questions before giving their consent. Participants will be informed that they have the right to withdraw their consent at any stage during the treatment.

Data protection and Participants' confidentiality

Queen's University Belfast carries the necessary and appropriate levels of indemnity for research involving human participants, giving cover for both negligent and non-negligent harm. It has policies and procedures that govern the collection, storage, quality assurance, and security of data. A Project Management Team, comprised of experienced co-investigators (CIs), will meet quarterly over the course of the study. They will assume responsibility for data integrity and quality.

QUB Research and Governance offices have robust processes for the oversight and governance of research, in particular, research involving human participants. All data used as part of this research will comply with all relevant legal requirements and codes of good practice. All QUB regulations relating to research involving human participants will be strictly adhered to and research staff will undertake the Good Clinical Practice training. All data will be anonymized, and participants' confidentiality maintained throughout. Participants will be allocated a unique ID Clinical colleagues in the Regional Trauma Network SET will be responsible for maintaining separate, confidential registers that will match each participant's unique ID with their name. These will be stored securely and separately from other data, with access limited to designated persons. Staff are required to read and follow the relevant security and data usage policies. All anonymized and pseudo anonymized data will be kept for five years, as per QUB Data management policy.

Paper files (consent forms) will be kept securely in locked filing cabinets in rooms requiring authenticated access in order to gain entry in SET. Interviews will be audio recorded and kept on an encrypted memory pen, transcribed verbatim stored securely within QUB grounds, and deleted within 2 weeks of recording. Access to data will be limited to designated staff only. All electronic data will be stored on password-protected computers. If participant(s) display signs of distress during or after interviews/focus groups (e.g., crying, or aggressive behavior), the researcher will report this to the RTN Clinical Lead/PI and follow the guidelines and protocols outlined by the organization.

It is worth noting that whilst the imagery and footage used to create personalized VR environments are specific to the participant's trauma, there will be no identifiable data within these. All imagery and footage will be saved and stored safely within the RTN and QUB research team.

Assessment and management of risk

The study will comply with the QUB and SET RTN risk policies. The clinical risk will be managed throughout the study by the clinicians who are delivering the treatment and the lead clinical research coordinator. SET trains the clinicians who are taking part in the study to manage patient-related risks and ensures that any risks that arise among participants are managed appropriately. They can manage the risk throughout the study. At the beginning of the study, a risk assessment will be conducted, and potential risk factors will be identified, i.e., risk of harm to self or others (e.g., expression of suicidal ideation), degree of distress associated with the problem, this is laid out in the RTN Screening Proforma. An agreed risk management plan with the participant will proceed throughout the study, a specific Distress Protocol has been designed for clinicians using the intervention in sessions and the follow-up interview held by the QUB Researcher at the end of the intervention. As Participants will be viewing images within a virtual environment specific to their traumatic experience, this may cause distress. Participants enrolled in the study will be allowed to contact clinicians should they become distressed in between weekly sessions and furthermore will receive advice from clinicians and be provided with contact information for services available to them should they have concerns regarding the safety of themselves or others, e.g., contacting their GP, accessing the Emergency Department. The potential risk concerning the use of VR apparatus will be managed via exclusion criteria, i.e., excluding high-risk medical conditions via health screening questions. So far, studies that used VR technology report no or minimal risk or adverse effects of participation, i.e., motion sickness, nausea, and headache. To minimize this temporary adverse effect and risk the investigators aim to keep VR exposure sessions within 30 minutes e.g., other studies have used 30-minute sessions and reported no risk and adverse reactions. Should any adverse effects or events take place during the treatment sessions, such as vomiting, reports of headaches, or neck pain, the clinician should record and report to the PI, who in turn will inform the QUB research team.

Infection Prevention and Control

The study will follow current SET guidelines regarding infection prevention and control. Participants will be advised to refrain from the study if they are experiencing any illnesses such as vomiting and/or diarrhea, coughs, colds, or flu-like symptoms and are demonstrating symptoms of any infectious conditions e.g., Covid-19, chicken pox, mumps, etc.

According to the updated Public Health Agency guidance, there is no longer a requirement for staff to wear masks in all Health and Social Care Settings. The use of fluid shield masks in patient-facing clinical areas should be determined on a risk assessment basis. Should the situation change, for example following the emergence of a new strain of COVID-19 giving cause for concern, then the study will follow update updated PHA guidance.

Prior to each visit participants will be advised to refrain from attending their treatment session at the RTN if they are experiencing the possible symptoms of COVID-19 (e.g., cough, fever, loss of smell or taste, fatigue), tested positive, or have been in contact with others who have Covid-19 symptoms.

Virtual Reality Headsets used in the study will be cleaned immediately after use.

Ethical And Regulatory Consideration

Below are some key ethical considerations and solutions related to the proposed study:

* All clinicians will be offered training sessions on the use of 360° video or VR Photoscan technology.
* Measures used at baseline will include validated scales and questions previously tested on PTSD patients and routinely used in clinical settings. All measures will be easy for participants to read and understand.
* Extra care will be taken to ensure participants understand the principle for informed consent and confidentiality as advised by good practice guidelines.
* A consent 'cooling-off' period approximately one week before the study is due to take place will take place.
* The research team and technical team will support clinicians.
* The clinicians will liaise with research staff to ensure that in so far as possible, individuals who are not suitable are removed from the study, e.g., underlying medical condition.
* Participants will not face disadvantages regardless of their decision to participate or withdraw from the study.
* The researchers will read and familiarise themselves with SET policies and procedures before conducting the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults who self-report the experience of type 1 trauma (NI related)
* PTSD symptoms as identified via PCL-5 > 31
* Ability to give informed consent
* Suitable and willingness to engage in TF-CBT
* Scene of the traumatic event is accessible for 360° video or VR Photoscan

Exclusion Criteria:

* History of severe motion sickness
* History of seizures, seizure disorder, or epilepsy
* History of bipolar disorder, psychosis, or schizophrenia
* Younger than 18 years old
* Experiences their trauma at a site that is not accessible (i.e., would not be possible to capture images)
* Previously engaged in TF-CBT within the PTS in the past 12 months
* Actively suicidal or undertaken suicidal action in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PCL 5 - Measure for PTSD | From enrolment to the end of treatment approx. week 16
  The PCL-5 is a 20 item self-report scale that assesses the 20 DSM-5 symptoms of PTSD and usually takes 5-10 minutes to complete. DSM-5 symptoms cluster severity scores can be obtained by summing the scores for the items within a given cluster i.e. Intrusion (5 items); avoidance (2 items); negative alteration in cognitions and mood (7 items) and alterations in arousal and reactivity (6 items). These items are rated on a 4-point Likert Scale ranging from 0 (not at all) to 4 (extremely) and are based on the participants experiences over the past month. Interpretation of the PCL-5 is made by the clinician and includes a total symptom severity score range 0-80 by summing the scores for each of the 20 items. A provisional PTSD diagnosis can be made using this scale and research suggests a PCL-5 cut off score between 31-33 is indicative of probable PTSD.
ITQ - International Trauma Questionnaire | From enrolment to the end of treatment approx. week 16
  The ITQ is an 18-question self-report measure that focuses on the core features of PTSD and Complex PTSD. All ITQ items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Scores are calculated for each symptom allowing clinicians to assess both PTSD and C-PTSD symptom severity. Higher scores typically indicate greater severity of trauma-related symptoms.

SECONDARY OUTCOMES:
Beck Depression Inventory-II | From enrolment to the end of treatment approx. week 16
  This tool is widely used to screen for depressive disorders and to measure the severity of depression. If appropriate, the clinician will administer at baseline and again post-therapy. The BDI-II includes 21 items, each of which corresponds to a symptom of depression and the maximum score is 63. For the BDI-II, a score of 10 to 18 indicates mild depression, and 30 or above indicates severe depression.
Igroup Presence Questionnaire | This measure will be given at the end of the first session where 360° video or VR Photoscan technology has been used. Approx. week 4
  IPQ is a subjective measure of presence in VR with high validity and internal consistency (α=.85) among virtual game players. The questionnaire includes 14 items rated on a 7-point Likert scale ranging from -3 (fully disagree) to +3 (fully agree) to measure a) spatial presence-a perception of being in the VR environment b) involvement-attention within the virtual environment and realness-how realistic the VR appears. Higher scores in a specific domain indicate a stronger presence.
Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) | From enrolment to the end of treatment approx. week 16
  CORE-OM make up a battery of self-report has 34 items designed to measure change due to psychological therapies and address wellbeing, problems, functioning and risk which takes approximately 10 minutes to complete. CORE-OM shows high internal consistency in clinical populations, all domains show appropriate internal validity i.e., α of >0.75 and <0.95. The items rated on a 5-point Likert scale ranging from 0 (not at all) and 5 (most or all of the time). In this study, CORE-OM will be used as another base line measure and taken again post treatment. Session by session outcome measures will also be taken and the shorter version CORE-10 which takes approximately 5 minutes to complete. This process (i.e., CORE-OM as base line measure and CORE-10 at each session) is recommended in research. Higher scores typically indicate greater impairment or worse outcomes.
Measurement of Subjective Unit of Distress Scale (SUDS) | This measure will be used during the sessions in which 360° video or VR Photoscan technology has been used. Approx. Week 4-8
  SUDS ratings are commonly used during exposure tasks in CBT for anxiety disorders. SUDS is used to indicate subjective perception of distress on a scale ranging from 0 (no distress) to 100 (extreme distress). During the VR sessions, clinicians will verbally ask clients their SUDS levels at 2-3 time points during the exposure. This will be recorded on a bespoke SUD's worksheet. At the end of the session, clinicians will also ask two short questions - 'Was there anything you liked about the VR experience? And was there anything you didn't like?
United Theory of Acceptance and Use of Technology (UTAUT2) Scale | Clinicians will complete a pre measure prior to enrolment and post, once they have completed the intervention using both arms of the technology. On average, one year.
  This measure is solely for the clinicians delivering the intervention. The UTAUT is a theoretical model developed to explain and predict the adoption and use of technology by individuals within organisations and other settings. It was created in 2003 and combines elements from several established technology acceptance theories. Scores range from 7 being the lowest and 35 being the highest. This model is often used in research to assess user attitudes and predict technology adoption in various fields, such as healthcare, education, and business. Higher scores in each of the constructs of the UTAUT model are generally considered better as they indicate positive perceptions and attitudes towards the technology.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Best, MSc in CBT, Principal Investigator — Queen's University, Belfast
Locations (1):
- South Eastern Health and Social Care Trust (Regional Trauma Network), Belfast, Dundonald, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study is part of a PhD project, and raw individual participant data will not be shared. However, anonymised results will be included in future publications to contribute to the broader research community.

REFERENCES:
- [Background] Rothbaum BO, Hodges LF, Ready D, Graap K, Alarcon RD. Virtual reality exposure therapy for Vietnam veterans with posttraumatic stress disorder. J Clin Psychiatry. 2001 Aug;62(8):617-22. doi: 10.4088/jcp.v62n0808. PMID 11561934
- [Background] Ehlers A, Clark DM, Hackmann A, McManus F, Fennell M. Cognitive therapy for post-traumatic stress disorder: development and evaluation. Behav Res Ther. 2005 Apr;43(4):413-31. doi: 10.1016/j.brat.2004.03.006. PMID 15701354
- [Background] Difede J, Hoffman H, Jaysinghe N. Innovative use of virtual reality technology in the treatment of PTSD in the aftermath of September 11. Psychiatr Serv. 2002 Sep;53(9):1083-5. doi: 10.1176/appi.ps.53.9.1083. No abstract available. PMID 12221305
- [Background] Blair C, Walsh C, Best P. Immersive 360 degrees videos in health and social care education: a scoping review. BMC Med Educ. 2021 Nov 24;21(1):590. doi: 10.1186/s12909-021-03013-y. PMID 34819063
- [Background] Beck JG, Coffey SF, Palyo SA, Gudmundsdottir B, Miller LM, Colder CR. Psychometric Properties of the Posttraumatic Cognitions Inventory (PTCI): a replication with motor vehicle accident survivors. Psychol Assess. 2004 Sep;16(3):289-98. doi: 10.1037/1040-3590.16.3.289. PMID 15456384
- [Background] Anderson PL, Price M, Edwards SM, Obasaju MA, Schmertz SK, Zimand E, Calamaras MR. Virtual reality exposure therapy for social anxiety disorder: a randomized controlled trial. J Consult Clin Psychol. 2013 Oct;81(5):751-60. doi: 10.1037/a0033559. Epub 2013 Jun 24. PMID 23796315
- [Background] Hess S, Zemishlany Z. [THE PSYCHIATRIC DIAGNOSIS GUIDE - DSM-5 - INNOVATIONS AND CRITICISM]. Harefuah. 2015 May;154(5):319-22, 338. Hebrew. PMID 26168644